CLINICAL TRIAL: NCT05726578
Title: Integrated Echocardiography and Chest Ultrasound Assessment of Lung Recruitment in Preterm Infants Using High Frequency Ventilation
Brief Title: Integrated Echocardiography and Chest Ultrasound Assessment of Lung Recruitment in Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0201752
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Ventilator Lung; Echocardiography; Chest Ultrasound; High Frequency Ventilation; Lung Recruitment
Keywords: Premature infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung recruitment (Experimental): preterm infants with moderate to severe respiratory distress
  Interventions: Other: Lung recruitment

INTERVENTIONS:
Other: Lung recruitment — establishment of lung recruitment using high frequency ventilation and assessment with chest ultrasound and echocardiography

SUMMARY:
The primary aim of this work is to evaluate the role of high frequency oscillatory ventilation (HFOV) in recruitment of lung in preterm newborns 32 to 37 weeks gestational age with moderate to severe respiratory distress. The secondary aim is to evaluate the role of chest ultrasound in monitoring of lung recruitment in comparison to routine chest x ray in those babies. Also cardiac hemodynamics will be assesed using functional echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Infants will be enrolled if they are 32 to 37 weeks of gestational age, have respiratory distress (RD) in the first 24 h of life, intubated and have invasive respiratory support using HFOV. Signs of RD are tachypnea (respiratory rate > 60/min), grunting, nasal flaring, chest retraction, and need of oxygen supplementation or other respiratory support.

Exclusion Criteria:

1. Known major congenital anomalies including congenital heart diseases.
2. Fetal hydrops.
3. Babies with congenital heart diseases

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
chest US | first 3 days after birth
  A mobile device (PHILIPS ® HD11 XE) with a 10-MHz linear probe will be used for chest ultrasound the 12 lung zones will be assessed regarding
  1. presence Of A lines, B-lines or C-profile
  2. presence or absence of pleural sliding
Superior Vena Cava flow in ml/kg/min | first 3 days of life
  Superior Vena Cava (SVC) Blood Flow using functional echocardiography
estimated pulmonary artery pressure in mmHg | first 3 days of life
  Pulmonary artery pressure (PAP) will be assessed by measuring tricuspid valve regurgitation peak velocity: this will be measured in apical 4 chamber view, with continous wave Doppler using modified Bernoulli equation. Systolic pulmonary artery pressure is equivalent to right ventricular systolic pressure in absence of outflow obstruction. Systolic Pulmonary Artery Pressure (SPAP) = Right Ventricular Systolic Pressure = 4x TR2 + Right Atrial Pressure (RAP), with RAP= 3-5 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hazem Wagih Gouda, PhD, Study Chair — Alexandria University; Ali Mohamed Abd Almohsen, PhD, Study Director — Alexandria University
Locations (2):
- Egypt (2):
  - Marwa Mohamed Farag, Alexandria
  - Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria